CLINICAL TRIAL: NCT00782548
Title: A Phase IV, Comparative, Randomized, Double Blind, Single-Dose, 2-way Crossover Study to Evaluate the Pharmacokinetics and Safety of Alpharma Branded Products Division (KADIAN)and Ligand Pharmaceuticals Inc. (Avinza) 30 mg Morphine Sulfate Sustained-Release Capsules in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Comparative Study to Evaluate KADIAN and Avinza in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Alan S. Marion, MD, PhD, MDS Pharma Services
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AA20003
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: KADIAN; morphine; Avinza; 30 mg; bioequivalence; fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Morphine; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Test product A (1 x 30 mg KADIAN)
  Interventions: Drug: KADIAN (morphine sulfate sustained-release) capsules
- 2 (Active Comparator): Reference product B (1 x 30 mg Avinza)
  Interventions: Drug: Avinza (morphine sulfate sustained-release) capsules

INTERVENTIONS:
Drug: KADIAN (morphine sulfate sustained-release) capsules — Capsules, 30 mg
  Other Names: Test product A
  Arms: 1
Drug: Avinza (morphine sulfate sustained-release) capsules — Capsules, 30 mg
  Other Names: Reference product B
  Arms: 2

SUMMARY:
The primary objective of this study was to compare the single-dose relative bioavailability of Alpharma Branded Products Division (Kadian®) and Ligand® Pharmaceuticals Inc. (AVINZA®) 30 mg morphine sulfate sustained-release capsules in healthy adult volunteers under fed conditions.

The secondary objective of this study was to evaluate the adverse events associated with each of these 2 different morphine sulfate modified-release commercial formulations

ELIGIBILITY:
Inclusion criteria:

* Healthy adult non-smoker, or moderate smokers (less than 10 cigarettes per day for at least 3 months) or ex-smoker (no smoking for at least 3 months) male or female volunteers, 19 to 40 years of age.
* Weighing at least 60 kg for males and 52 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983).
* Medically healthy subjects with no clinically significant abnormalities in their laboratory profile and ECGs, as deemed by the Principal Investigator.
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

  1. surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum.
  2. IUD in place for at least 3 months;
  3. barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study;
  4. surgical sterilization of the partner (vasectomy for 6 months minimum);
  5. hormonal contraceptives for at least 3 months prior to the first dose of the study.

Other birth control methods may have been deemed acceptable. Postmenopausal women with amenorrhea for > than 2 year, and confirmed by blood testing.

* Voluntarily consent to participate in the study.

Exclusion criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  1. alcoholism or drug abuse within the past 2 years;
  2. asthma or other chronic respiratory illness;
  3. gastrointestinal dysmobility or recent enteritis;
  4. hypersensitivity or idiosyncratic reaction to morphine or other opioids;
  5. hypersensitivity or idiosyncratic reaction to naltrexone, naloxone, or other narcotic antagonists.
* Female subjects who were pregnant or lactating.
* Subjects who had a surgery of the gastrointestinal tract (except appendectomy) which would interfere with absorption of the study drug
* Subjects who received hepatic enzyme inducing drugs (e.g. Nizoral®, Tagamet®) within the previous three months
* Subjects whose sitting blood pressure was less than 110/60 mm Hg at screening or 100/55 mm Hg before dosing.
* Subjects who were on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who had made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 56 days prior to the study.
* Subjects who had made a plasma donation within 7 days prior to the study.
* Subjects with hemoglobin less than 12.0 g/dL.
* Subjects who had participated in another clinical trial within 28 days prior to the first dose.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Plasma samples analyzed for morphine, morphine-3-glucuronide, and morphine-6-glucuronide | 60 hours post-dose

SECONDARY OUTCOMES:
To evaluate the adverse events associated with each of these 2 different morphine sulfate modified-release commercial formulations | monitored throughout study, until resolution

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Marion, MD, PhD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States